CLINICAL TRIAL: NCT03563170
Title: Molecularly Informed Integrated Immunotherapy Combining Innate High-affinity Natural Killer (haNK) Cell Therapy w/ Adenoviral & Yeast-based Vaccines to Induce T-cell Responses in Subjects w/ Advanced, Unresectable & Untransplantable HCC
Brief Title: QUILT-3.072: NANT Hepatocellular Carcinoma (HCC) Vaccine
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment not initiated
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.072
Record Dates: First submitted 2018-05-22; First posted 2018-06-20 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Hepatocellular Carcinoma Recurrent
Keywords: HCC
MeSH Terms: interventions — avelumab; Capecitabine; Cyclophosphamide; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Sorafenib; yeast-CEA vaccine; Cetuximab; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NANT Hepatocellular Carcinoma Vaccine (Experimental): Phase 1b and 2: The following combination of agents will be administered to subjects assigned to this treatment: Aldoxorubicin HCl, ETBX-011, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, N-803, haNK™, avelumab, capecitabine, cetuximab, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, sorafenib tosylate, SBRT.
  Interventions: Biological: ETBX-011; Biological: GI-4000; Biological: haNK for infusion; Biological: avelumab; Drug: Capecitabine; Drug: Cyclophosphamide; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: nab-Paclitaxel; Drug: Sorafenib; Procedure: SBRT; Biological: Aldoxorubicin hydrochloride; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-6207; Biological: GI-6301; Drug: Cetuximab; Biological: N-803
- Sorafenib Monotherapy (Active Comparator): Phase 2: Sorafenib monotherapy will be administered to subjects with advanced, unresectable, and untransplantable HCC, who have not previously received sorafenib, and who are randomly assigned to receive SOC treatment.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: GI-4000 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant RAS proteins
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: haNK for infusion — NK-92 [CD16.158V, ER IL-2]
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: avelumab — Recombinant human anti-PD-L1 IgG1 monoclonal antibody
  Arms: NANT Hepatocellular Carcinoma Vaccine
Drug: Capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
  Arms: NANT Hepatocellular Carcinoma Vaccine
Drug: Cyclophosphamide — anhydrous
  Arms: NANT Hepatocellular Carcinoma Vaccine
Drug: 5-Fluorouracil — 5-FU; Fluorouracil
  Arms: NANT Hepatocellular Carcinoma Vaccine
Drug: Leucovorin — Leucovorin calcium salt
  Arms: NANT Hepatocellular Carcinoma Vaccine
Drug: nab-Paclitaxel — ABRAXANE® [paclitaxel protein-bound particles for injectable suspension] [albumin-bound]
  Arms: NANT Hepatocellular Carcinoma Vaccine
Drug: Sorafenib — NEXAVAR® tablets, for oral use
Procedure: SBRT — Stereotactic Body Radiation Therapy
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: Aldoxorubicin hydrochloride — HCl
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury vaccine
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: ETBX-061 — Ad5 [E1-, E2b-]-mucin 1 [MUC1] vaccine
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: GI-6207 — CEA yeast vaccine
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: GI-6301 — Brachyury yeast vaccine
  Arms: NANT Hepatocellular Carcinoma Vaccine
Drug: Cetuximab — ERBITUX® injection, for IV infusion)
  Arms: NANT Hepatocellular Carcinoma Vaccine
Biological: N-803 — Recombinant human super agonist IL-15 complex [also known as IL-15N72D:IL- 15RαSu/IgG1 Fc complex]
  Arms: NANT Hepatocellular Carcinoma Vaccine

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with advanced, unresectable, and untransplantable HCC.

DETAILED DESCRIPTION:
Treatment will be administered in two phases, an induction and a maintenance phase. Subjects will continue induction treatment for up to 1 year. Those who have a CR in the induction phase will enter the maintenance phase of the study. Subjects who experience ongoing SD or an ongoing PR at 1 year may enter the maintenance phase at the Investigator's and Sponsor's discretion. Subjects may remain in the maintenance phase of the study for up to 1 year. Treatment in the study will be discontinued if the subject experiences confirmed PD or unacceptable toxicity (not corrected with dose reduction), withdraws consent, undergoes liver transplantation or surgical resection, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. Subjects with an initial assessment of PD may, at the discretion of the Investigator, continue to receive study treatment until PD is confirmed. The maximum time on study treatment is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed advanced, unresectable and untransplantable HCC.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. Must have Child-Pugh class A only.
7. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen following the conclusion of the most recent anticancer treatment and be willing to release the specimen for prospective and exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
8. Must be willing to provide blood samples prior to the start of treatment on this study for prospective tumor molecular profiling and exploratory analyses.
9. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment for exploratory analyses, if considered safe by the Investigator.
10. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
11. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.
12. Any prior locoregional therapy allowed.

    Phase 1b only
13. Must have progressed or experienced unacceptable toxicity on sorafenib prior to enrollment in the study.

    Phase 2 single-arm component only
14. Must have progressed on or after sorafenib monotherapy in the randomized phase 2 portion of the study OR progressed or experienced unacceptable toxicity on sorafenib prior to enrollment on the study.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, or autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count < 1,000 cells/mm^3
   2. Medically uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
   3. Platelet count < 75,000 cells/mm^3.
   4. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   5. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT])

      ≥ 2.5 × ULN (≥ 5 × ULN in subjects with liver metastases).
   6. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   8. International normalized ratio (INR) ≥ 2.0
   9. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
7. Episode of portal hypertension-related GI bleeding within prior 6 months.
8. Serious myocardial dysfunction defined by echocardiogram (ECHO) as absolute left ventricular ejection fraction (LVEF) 10% below the institution's lower limit of normal (LLN).
9. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
10. Positive results of screening test for human immunodeficiency virus (HIV).
11. Participants with dual active hepatitis B virus (HBV) infection (hepatitis B surface antigen [HBsAg] positive [+] and /or detectable HBVDNA) and hepatitis C virus (HCV) infection (anti-HCV antibody [Ab] [+] and detectable HCV ribonucleic acid [RNA]) at study entry. Subjects with chronic infection by HCV who are treated with anti-hepatitis B therapy (successfully or treatment failure) or untreated are allowed on study. Controlled (treated) hepatitis B subjects will be allowed if they meet the following criteria:

    1. Antiviral therapy for HBV must be given for at least 12 weeks and HBV viral load must be less than 100 IU/mL prior to first dose of study drug; subjects on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study treatment.
    2. Subjects who are positive for anti-hepatitis B core Abs (HBc[+]), negative for HBsAg, negative for anti-hepatitis B surface Ab (HBs[-]), and have a HBV viral load under 100 IU/mL do not require HBV anti-viral prophylaxis.
    3. Subjects with successful HCV treatment are allowed as long as there are at least 4 weeks between achieving sustained viral response (SVR) and start of study drug.
12. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
13. Known hypersensitivity to any component of the study medication(s).
14. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
15. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
16. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
17. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
18. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
19. Concurrent participation in any interventional clinical trial.
20. Pregnant and nursing women.

    Phase 2 randomized component only -
21. Prior sorafenib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs and SAEs, graded using the NCI CTCAE Version 4.03 | 2 years
  Phase 1b
Evaluate the overall safety profile in subjects with advanced, unresectable, untransplantable HCC who have progressed or experienced unacceptable toxicity on prior sorafenib treatment. Measured / reported based on the tumor size imaging per RECIST 1.1. | 2 years
  Phase 1b
Progression Free Survival from baseline to progression, per RECIST 1.1 | 2 years
  Phase 2 Randomized Component
Overall Response Rate, as determined by the percentage of patients achieving Partial or Complete Response per RECIST 1.1 | 2 years
  Phase 2 Single Arm Component

SECONDARY OUTCOMES:
ORR for Phase 1b and Phase 2 Randomized Component | 2 years
  Overall Response Rate, as determined by the percentage of patients achieving Partial or Complete response per RECIST 1.1 and irRC
PFS for Phase 1b and Phase 2 Single Arm Component | 1 year
  Progression Free Survival from baseline to progression per RECIST 1.1 and irRC
OS for Phase 1b, Phase 2 Randomized, and Phase 2 Single Arm Component | 2 years
  Overall Survival from first treatment to date of death (any cause)
DOR for Phase 1b, Phase 2 Randomized, and Phase 2 Single Arm Component | 2 years
  Duration of Response from date of first response to date of disease progression or death (any cause), per RECIST 1.1 and irRC
DCR for Phase 1b, Phase 2 Randomized, and Phase 2 Single Arm Component | 1 year
  Disease Control Rate: the number of patients with a CR, PR or SD lasting at least 2 months per RECIST 1.1 and irRC
QoL for Phase 1b, Phase 2 Randomized, and Phase 2 Single Arm Component | 1 year
  Quality of Life as assessed by Patient Reported Outcomes using the FACT-C questionnaire
PFS for Phase 2 Randomized Component | 2 years
  Progression Free Survival from baseline to progression per irRC
Safety for Phase 2 Randomized and Single Arm Component | 2 years
  Incidence of treatment-emergent AEs and SAEs, graded using the NCI CTCAE Version 4.03
ORR for Phase 2 Single Arm Component | 2 years
  Overall Response Rate, as determined by the percentage of patients achieving Partial or Complete response per irRC

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States